CLINICAL TRIAL: NCT06552429
Title: A Phase 2 Multicenter, Randomized, Open-label Study to Evaluate the Pharmacokinetic, Safety and Efficacy of Peginterferon Alfa-2b Injection in Subjects With Essential Thrombocythemia Who Are Resistant to or Intolerant of Hydroxyurea.
Brief Title: Peginterferon α-2b Injection for Hydroxyurea Resistant or Intolerant ET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2b-4-3-002
Record Dates: First submitted 2024-07-27; First posted 2024-08-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Essential Thrombocythemia
Keywords: Essential Thrombocythemia; Peginterferon α-2b; hydroxyurea resistant; hydroxyurea intolerant
MeSH Terms: conditions — Thrombocythemia, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peginterferon α-2b 135 mcg dose group (Experimental)
  Interventions: Drug: Peginterferon α-2b injection
- Peginterferon α-2b 180 mcg dose group (Experimental)
  Interventions: Drug: Peginterferon α-2b injection

INTERVENTIONS:
Drug: Peginterferon α-2b injection — Peginterferon α-2b injection, 135 mcg, s.c., once a week, during the targeted treatment period (the first 48 week), peginterferon α-2b dose is depended on the patient's response and tolerability during the extension treatment (week 49 to week 96).
  Arms: Peginterferon α-2b 135 mcg dose group
Drug: Peginterferon α-2b injection — Peginterferon α-2b injection, 180 mcg, s.c., once a week, during the targeted treatment period (the first 48 week), peginterferon α-2b dose is depended on the patient's response and tolerability during the extension treatment (week 49 to week 96).
  Arms: Peginterferon α-2b 180 mcg dose group

SUMMARY:
This is a multicenter, randomized, open-label Phase 2 clinical study. It is aimed to enroll 27 essential thrombocytopenia (ET) patients who are resistant to or intolerant of hydroxyurea(HU). Eligible patients will be randomized to receive either Peginterferon α-2b 135 mcg or Peginterferon α-2b 180 mcg at a ratio of 1:2, and all subjects will go through a target treatment period (Weeks 1 ~ Week 48), an extension treatment period (Weeks 49 ~ Week 96) and a follow-up period (Weeks 97 ~ Week 100). Pharmacokinetics, safety, efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged greater or equal to 18 years old at screening;
* Subjects diagnosed as high-risk ET according to the World Health Organization (WHO) 2016 criteria：1) who is older than 60 years and JAK2V617F positive at screening, 2) or who previously suffered from disease-related thrombosis or hemorrhage;
* Subjects who have previously received HU for ET, and the time interval between the last HU dose and the first dose of the study drug should not be less than 7 days;
* Interferon treatment-naïve, and for those who have previously received interferon the the time interval between the last dose of interferon and randomization should not be less than 1 month;
* Patients with confirmed hydroxyurea resistance or intolerant, as at least one of the following criteria is met:

  1. Platelet count remain greater than 600×10^9 /L after at least 3 months of HU treatment at a dose ≥2g/d (dose ≥2.5 g/d if subject weight > 80 kg);
  2. Platelet count greater than 400*10^9/L while white blood cell (WBC) count lower than 2.5*10^9/L, or platelet count greater than 400*10^9 /L while hemoglobin lower than 100 g/L at any dose of HU;
  3. Presence of HU-related toxicities at any dose of HU: e.g. ulcers in legs, or any unacceptable skin mucosal manifestations or fever;
* Platelet counts > 450*10^9/L at screening;
* Neutrophil count ≥1.0*10^9/L at screening;
* Haemoglobin ≥11 g/dL at screening for males and 10 g/dL for females at screening;
* There is no serious function damage in liver and kidney: total bilirubin ≤1.5 upper limit of normal (ULN), alanine aminotransferase≤2.0 ULN, aspartate aminotransferase≤2.0 ULN, prothrombin time is prolonged by less than 4 seconds, Creatinine clearance ≥50 mL/min (according to Cockcroft-Gault formula) at screening;
* Both male and female subjects must agree take an appropriate contraceptive method, including:

  1. Male subjects: must agree to use reliable contraception from inform consent until 6 months following the last dose of the study drug.
  2. Female subjects: Must meet at least one of the following conditions:

  i) Women without childbearing potential; ii) Women of childbearing potential: no pregnant or breastfeed, negative in blood pregnancy test within 4 days prior to the first dosing, and must agree to use reliable contraception from inform consent until 6 months following the last dose of the study drug;
* Subjects understand the objective, characteristic, method and possible adverse reactions of the study, voluntarily participate in this study, and sign informed consent.

Exclusion Criteria:

* History of any other myeloproliferative tumors, or evidence of the presence of any other myeloproliferative tumors;
* Contraindications or hypersensitivities to interferons of any of its excipients;
* Severe medical conditions or serious comorbidities that the investigators determined could jeopardize the safety or protocol adherence, e.g. New York Heart Association [NYHA] Class III-IV, congestive heart failure, symptomatic arrhythmias，pulmonary hypertension;
* History of major organ transplantation;
* Documented autoimmune disease or history of autoimmune disease at screening, e.g. medication un-controlled thyroid dysfunction, autoimmune hepatitis, idiopathic thrombocytopenic purpura, scleroderma, psoriasis, or any autoimmune arthritis;
* Clinically significant pulmonary infiltration, infectious pneumonia, and non-infectious pneumonia at screening that, in the investigator's opinion, would jeopardize the safety of the subject or their compliance with the protocol;
* Infection with systemic clinical manifestations at screening, e.g., bacteria, fungi, human immunodeficiency virus, excluding hepatitis B and/or C;
* Evidence of severe retinopathy, e.g., cytomegalovirus retinitis, symptomatic macular degeneration, or clinically significant eye disease, e.g. due to diabetes mellitus or hypertension;
* Diagnosed clinically significant depression or a history of depression and, in the investigator's opinion, previous suicide attempts or at any risk of suicide at screening;
* Diagnosed clinically significant neurological disease or a history of clinically significant neurological disease, except for a history of stable cerebral thrombosis or cerebral hemorrhage;
* History of any malignancy within 5 years (except stage 0 chronic lymphocytic leukemia, basal cell carcinoma, squamous cell carcinoma, and superficial melanoma);
* A history of alcohol or drug abuse within 1 year;
* Have used any investigational drug within 4 weeks prior to first dose of investigational drug, or not recovered from the effects of prior investigational drug administration;
* Other situations that, in the investigator's opinion, not appropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-10-26 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | week1,4, 8, 12, 24, 36, 48, 60, 72, 84, 96.
Time to maximum concentration (Tmax) | week1,4, 8, 12, 24, 36, 48, 60, 72, 84, 96.
Area under the plasma concentration-time curve | week1,4, 8, 12, 24, 36, 48, 60, 72, 84, 96.
Apparent volume of distribution after oral administration (Vz/f) | week1,4, 8, 12, 24, 36, 48, 60, 72, 84, 96.
Apparent plasma clearance (CL/F) | week1,4, 8, 12, 24, 36, 48, 60, 72, 84, 96.
Plasma elimination half-life (t1/2) | week1,4, 8, 12, 24, 36, 48, 60, 72, 84, 96.
Relationship between exposure and the effect (desired-effectiveness or undesirable-toxicity) in a pharmacokinetic model and pharmacodynamic model. | up to 96 weeks.

SECONDARY OUTCOMES:
Rate of complete hematological remission. | Week 24, 36, 48, 60, 72, 84, 96.
Platelet counts change from baseline. | Week 12, 24, 36, 48, 60, 72, 84, 96.
White blood cell counts change from baseline. | Week 12, 24, 36, 48, 60, 72, 84, 96.
Complete remission rate. | Week 24, 36, 48, 60, 72, 84, 96.
Time to complete remission from baseline. | Week 48, 96.
Duration of complete remission. | Week 48, 96.
Remission rate of bone marrow. | Week 48, 96.
Incidence of disease progression. | Week 48, 96.
Change of JAK2V617F mutations load from baseline. | Week 48, 96.
  JAK2V617F mutations were quantitatively detected using next-generation sequencing
Change of CALR mutations load from baseline. | Week 48, 96.
  CALR mutations were quantitatively detected using next-generation sequencing
Change of MPL mutations load from baseline. | Week 48, 96.
  MPL mutations were quantitatively detected using next-generation sequencing
Change of MPN-SAF TSS scores from baseline | Week 12, 24, 36, 48, 60, 72, 84,96.
Change of spleen size from baseline | Week 12, 24, 36, 48, 60, 72, 84, 96.
  The maximum length of the spleen was measured by ultrasound.
Rate of complete hematological remission maintenance in patients received dose-reduction extension therapy | Week 96.
Duration of complete hematological remission in patients received dose-reduction extension therapy | Week 96.
Change of 3-level Version of EuroQol Five Dimensions(EQ-5D-3L) scores from baseline. | Week 12, 24, 36, 48, 60, 72, 84, 96.
Incidence of thrombotic and bleeding events. | through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Principal Investigator — Chinese Academy of Medical Sciences
Locations (8):
- China (8):
  - Peking Union Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University People's Hospital, Beijing
  - Union Hospital affiliated to Fujian Medical University, Fujian
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Harbin First Hospital, Harbin
  - Henan Cancer Hospital, Henan
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang

IPD SHARING:
Plan to Share IPD: No